CLINICAL TRIAL: NCT01572558
Title: Conservative Treatment of Acute Appendicitis in Children Pilot Trial
Brief Title: Conservative Treatment of Acute Appendicitis in Children
Acronym: CONSAPP Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jan Svensson, Principal investigator, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA2011/4:8
Record Dates: First submitted 2012-02-13; First posted 2012-04-06 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Appendicitis; Child
Keywords: Appendectomy; Nonsurgical treatment with antibiotics
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy; Meropenem; Metronidazole; Benchmarking; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Appendectomy (Active Comparator): Standard surgical treatment, appendectomy
  Interventions: Procedure: Appendectomy
- Conservative, non-surgical treatment (Experimental): Non-operative treatment with intravenous and oral antibiotics
  Interventions: Drug: Conservative, non-surgical treatment

INTERVENTIONS:
Procedure: Appendectomy — Standard surgical treatment, normally laparoscopic appendectomy
  Other Names: Open appendectomy; Laparoscopic appendectomy
  Arms: Appendectomy
Drug: Conservative, non-surgical treatment — Non-surgical treatment, intravenous and oral antibiotics. Meropenem and Metronidazol will be used as intravenous antibiotics, Ciprofloxacin and Metronidazol will be used as oral antibiotics.
  Other Names: Meronem®; Meropenem; Flagyl®; Metronidazol; Ciproxin®; Ciprofloxacin
  Arms: Conservative, non-surgical treatment

SUMMARY:
This is a feasibility study that will be performed at the Astrid Lindgren Children´s Hospital, Karolinska University Hospital, Stockholm, Sweden. It will involve 50 patients, randomized to either conservative, non-operative, treatment with antibiotics OR surgery. The study will test an computerized randomization system, the availability of patients willing to participate in the trial and the trial protocol. The investigators will assess the characteristics of the patients who agree to participate in the study and those who do not. The investigators will explore short term outcome and design suitable long term outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Children 5-15 years old with a clinical diagnosis of appendicitis that prior to the trial would have been subjected to a surgical intervention

Exclusion Criteria:

* Suspicion of perforated appendicitis on the basis of generalized peritonitis
* An appendiceal mass, diagnosed either by palpation or with radiology

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Resolution of symptoms without significant complications | 30 days
  This outcome measure is designed to be similar between the two groups. It is measured in number of participants that fails its designated treatment.
  Failure of treatment include abscess formation requiring treatment (prolonged antibiotic course or drainage), wound infection requiring intravenous antibiotics, wound dehiscence requiring treatment, prolonged ileus >5 days, length of stay >7 days, recurrent appendicitis, persistance of symptoms leading to surgery and negative appendectomy.

SECONDARY OUTCOMES:
Time in hospital | 7 days
  Number of days as inpatients after initiation of allocated treatment, ea. after randomization.
Time to resolution of symptoms | 7 days
  In hours, to the time where there is no significant pain (VAS not more than 3), no temprature nor any anorexia.
Abscess formation | 7 days
  As noted either in hospital or during follow up.
Early complications | 7 days
  Wound infections, wound dehiscence, diarrhea etc.
Pain | 48 hours
  Measured after 12, 24 and 48 hours with the 0-10 Visual Analoge Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jan F Svensson, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Astrid Lindgren Children´s Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Patkova B, Svenningsson A, Almstrom M, Eaton S, Wester T, Svensson JF. Nonoperative Treatment Versus Appendectomy for Acute Nonperforated Appendicitis in Children: Five-year Follow Up of a Randomized Controlled Pilot Trial. Ann Surg. 2020 Jun;271(6):1030-1035. doi: 10.1097/SLA.0000000000003646. PMID 31800496
- [Derived] Svensson JF, Patkova B, Almstrom M, Naji H, Hall NJ, Eaton S, Pierro A, Wester T. Nonoperative treatment with antibiotics versus surgery for acute nonperforated appendicitis in children: a pilot randomized controlled trial. Ann Surg. 2015 Jan;261(1):67-71. doi: 10.1097/SLA.0000000000000835. PMID 25072441